CLINICAL TRIAL: NCT03428789
Title: Sensory Recovery of the Breast Following Innervated and Non-innervated DIEP Flap Breast Reconstructions
Brief Title: Nerve Coaptation in DIEP Flap Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Rene van der Hulst, Prof. Dr., Maastricht University Medical Center
Other Study IDs: METC 16-4-147
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: breast reconstruction; DIEP flap; Nerve coaptation; Sensory recovery
MeSH Terms: conditions — Breast Neoplasms | interventions — Nerve Transfer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Innervated DIEP flaps: Patients in this group underwent immediate or delayed, unilateral or bilateral deep inferior epigastric artery perforator (DIEP) flap breast reconstruction with additional sensory nerve coaptation.
  Interventions: Procedure: Sensory nerve coaptation
- Non-innervated DIEP flaps: Patients in this group underwent immediate or delayed, unilateral or bilateral deep inferior epigastric artery perforator (DIEP) flap breast reconstruction without sensory nerve coaptation.

INTERVENTIONS:
Procedure: Sensory nerve coaptation — A recipient sensory nerve of the abdomen was reattached to a donor nerve in the chest area. The sensory branch of usually the 11th intercostal nerve was used as recipient nerve for nerve coaptation and the anterior cutaneous branch of the third intercostal nerve was used as donor nerve. Direct, end-to-end nerve coaptation was performed with two stitches.
  Other Names: Neurotization; Neurorrhaphy; Reinnervation
  Groups: Innervated DIEP flaps

SUMMARY:
The sensory recovery of the breast remains an undervalued aspect of breast reconstruction and surgical reinnervation is not regarded as a priority by most reconstructive surgeons. A prospective study was conducted of all patients who underwent either innervated or non-innervated DIEP flap breast reconstruction in Maastricht University Medical Center and returned for follow-up between September 2015 and July 2017. Semmes-Weinstein monofilaments were used for sensory testing of the breast. This study showed that nerve coaptation in DIEP flap breast reconstruction resulted in a significantly improved sensation of the reconstructed breast compared to non-innervated flaps.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years or older
* Unilateral or bilateral DIEP flap breast reconstruction
* Returned for follow-up between September 2015 and July 2017
* Informed consent

Exclusion Criteria:

* Bilateral breast reconstruction with a unilateral innervated DIEP flap and a contralateral non-innervated flap
* Flaps that required a take-back

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients of 18 years or older.
Study Population: In this prospective study, patients who underwent an innervated or non-innervated DIEP flap breast reconstruction between January 2010 and July 2016 at Maastricht University Medical Center in the Netherlands were included if they returned for follow-up between September 2015 and July 2017.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
The extent of sensory recovery of the reconstructed breast to touch | Through study completion up to 24 months postoperatively
  The sensory recovery of the breast to touch was tested at different follow-up moments after the initial surgery. Semmes-Weinstein monofilaments were used for sensory testing. Nine areas of the breast, indicating native skin and flap skin, were tested. Mean monofilament values were calculated for each area and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: René van der Hulst, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No